CLINICAL TRIAL: NCT04509882
Title: Add-on Study of Bear Bile Pill for Patients With Major Depressive Disorder (MDD)
Brief Title: Bear Bile Pill as add-on the Treatment of MDD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Jingjing HUANG, Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCTNCT04002259
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bear bile pill (Experimental): Patients randomized to the bear bile pill arm will receive treatment with 15 pills, three times daily of bear bile pill (1350mg per day) plus on-going antidepressant therapy (SSRI/SNRI).
  Interventions: Drug: bear bile pill
- placebo (Placebo Comparator): Patients randomized to the placebo arm will receive 15 pills, three times daily of placebo plus on-going antidepressant therapy (SSRI/SNRI).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bear bile pill — Bear bile pill (15 pills) taken orally three times a day after meals with water.
  Arms: bear bile pill
Drug: placebo — Placebo(15 pills) taken orally three times a day after meals with water.
  Arms: placebo

SUMMARY:
This is a single-center, double blind, randomized, placebo-controlled, parallel group study of bear bile pill, as add-on therapy in MDD patients conducted in Shang Hai Mental Health Center. The purpose of this study is to determine the efficacy and safety of bear bile pill in reducing symptoms of depression in Major Depressive Disorder (MDD)patients with inadequate response to current antidepressant therapy. Following a screening period, subjects who meet the entry criteria will be randomized to treated with either placebo or 450mg bear bile pill three times daily for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the Diagnostic and Statistical Manual of Mental Disorder, Fifth Edition, Text Revision (DSM-V) criteria for Major Depressive Disorder (MDD); a single or recurrent episode without psychotic features ;Codes are as follows: F32.0、F32.1、F32.2、F33.0、F33.1 、F33.2.
2. Outpatients or inpatients.
3. Male or female subjects aged 18-65 years.
4. Patients have got standard treatment of SSRI/SNRI monotherapy for more than 4 weeks in current episode of depression before trial entry.
5. MADRS score greater than 20.
6. Women of childbearing potential must be willing to use acceptable methods of contraception throughout the study period and the following one month.
7. The patient the patient fully understand and signed the informed consent form

Exclusion Criteria:

1. Patient has survived a suicide attempt or has acute suicidal tendencies (MADRS Item 10 > 4).
2. Comorbidity according to DSM-V, axis I except major depressive disorder.
3. Failed 3 or more adequate antidepressant courses in current episode of depression.
4. MADRS reduction ratio ≥25% within one week from the screening to the baseline Visit.
5. Depressive episode secondary to psychiatric illness or somatic disease.
6. Serious and instable body disease such as cerebrovascular disease, liver and kidney disease, disease of internal secretion (abnormal thyroid function), blood disease; any history of seizures or other organic brain diseases.
7. History of alcohol or drug abuse over the last 6 months
8. Allergic history to bear bile pills, or serious drug allergic history.
9. Pregnant or lactating women and women of childbearing potential throughout the study period; men who have the desire of fertility within six months;
10. Clinically significant changes in ECG or laboratory tests, including >1.5X upper limit of normal liver function、over the limit of normal renal function and blood sugar、abnormal cardiac troponins、obvious abnormity in the thyroid function
11. Treatment with MECT or rTMS in nearly three months.
12. Treatment with a systematic psychological treatment in nearly three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in the total Montgomery-Asberg Depression Rating Scale (MADRS) score between randomization and end of study. | assessed from baseline to week 8(end of study)
  The main objective is to explore whether bear bile pill add on SSRI or SNRI will improve the MDD symptoms after 8 weeks of treatment, and investigators assess the scale at baseline and week 1, 2, 4, 8.

SECONDARY OUTCOMES:
Effective treatment | assessed from baseline to week 8 (end of study)
  effectivity：MADRS or HAMD reduction ratio ≥50% reductive ratio: [（Baseline score- Endpoint score）／Baseline score]×100%
Clinical remission rate | assessed from baseline to week 8 (end of study)
  patients who are in remission at the end of the study will be summarized by treatment group, MADRS score ≤12 or HAMD-17≤7.
The Montgomery-Asberg Depression Rating Scale (MADRS) reduction ratio | assessed from baseline to week 8 (end of study)
  MADRS reduction ratio were used to evaluate the effectiveness of the treatment,and investigators assess the scale at baseline and week 1, 2, 4, 8.
The Hamilton Depression Rating Scale (HAM-D17) reduction ratio | assessed from baseline to week 8 (end of study)
  the Hamilton Depression Rating Scale reduction ratio were used to evaluate the effectiveness of the treatment,and investigators assess the scale at baseline and week 1, 2, 4, 8.
change in the total score of the Hamilton Anxiety Scale(HAMA) | assessed from baseline to week 8 (end of study)
change in total score of the Clinical Global Impression-Severity (CGI-S) scale. | assessed from baseline to week 8 (end of study)
change in total score of the Clinical Global Impression-Improvement (CGI-I) scale. | assessed from baseline to week 8 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing huang, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Jing jing Huang, Shanghai, China